CLINICAL TRIAL: NCT00024050
Title: Allogeneic Peripheral Blood Stem Cell (PBSC) Transplantation for the Treatment of "Less Advanced" Myelodysplasi
Brief Title: Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Myelodysplastic Syndrome
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: 1536.00; FHCRC-1536.00; NCI-G01-2009; CDR0000068887 (Registry Identifier: PDQ)
Record Dates: First submitted 2001-09-13; First posted 2003-01-27 (Estimated); Last update posted 2010-05-13 (Estimated); Status verified 2010-05

CONDITIONS: Leukemia; Myelodysplastic Syndromes
Keywords: refractory anemia; refractory anemia with ringed sideroblasts; de novo myelodysplastic syndromes; previously treated myelodysplastic syndromes; secondary myelodysplastic syndromes; childhood myelodysplastic syndromes
MeSH Terms: conditions — Leukemia; Myelodysplastic Syndromes; Anemia, Refractory | interventions — Busulfan; Cyclophosphamide; Cyclosporine; Methotrexate; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: methotrexate
Procedure: allogeneic bone marrow transplantation
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy.

PURPOSE: Phase II trial to study the effectiveness of chemotherapy followed by peripheral stem cell transplantation in treating patients who have myelodysplastic syndrome.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the non-relapse toxicity and mortality on day 100 and at 1 year after transplantation in patients with low or intermediate-risk myelodysplastic syndrome treated with busulfan, cyclophosphamide, and allogeneic peripheral blood stem cell transplantation.
* Determine the incidence of donor stem cell engraftment and relapse-free survival in these patients treated with this regimen.
* Determine the incidence and severity of acute and chronic graft-versus-host disease and invasive fungal infections in these patients treated with this regimen.
* Determine the incidence of relapse in these patients treated with this regimen.

OUTLINE: Peripheral blood stem cells (PBSC) or bone marrow are harvested from a related or unrelated compatible donor. PBSC are selected for CD34+ cells.

Patients receive oral busulfan every 6 hours on days -7 to -4 and cyclophosphamide IV on days -3 and -2. Allogeneic PBSC or bone marrow is infused on day 0.

As graft-versus-host disease prophylaxis, patients receive cyclosporine IV beginning on day -1 and continuing orally twice daily (if feasible) until day 51 followed by a taper. Patients also receive methotrexate IV on days 1, 3, 6, and 11.

Patients are followed through day 100, every 6 months for 2 years, and then annually thereafter.

PROJECTED ACCRUAL: A total of 40 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of low or intermediate-risk myelodysplastic syndrome

  * Refractory anemia (RA)
  * RA with ringed sideroblasts
* No advanced myelodysplastic syndrome (i.e., at least 5% blasts in the marrow, more than 1% blasts in the peripheral blood, or blasts in the cerebrospinal fluid)
* No poor-risk cytogenetics (i.e., abnormalities of chromosome 7 or complex abnormalities)
* HLA-A, B, C, DRB1, and DQB1 compatible related or unrelated donor available

  * Mismatch for a single HLA-A, B, C, DRB1, or DQB1 allele allowed

PATIENT CHARACTERISTICS:

Age:

* 65 and under

Performance status:

* Not specified

Life expectancy:

* Not specified

Hematopoietic:

* Not specified

Hepatic:

* AST no greater than 2 times normal

Renal:

* Creatinine no greater than 2 times upper limit of normal
* Creatinine clearance at least 50%

Cardiovascular:

* No cardiac insufficiency requiring treatment
* No symptomatic coronary artery disease

Pulmonary:

* No severe hypoxemia (pO2 less than 70 mm Hg with DLCO less than 70% predicted)
* No mild hypoxemia (pO2 less than 80 mm Hg with DLCO less than 60% predicted)

Other:

* No other disease that would limit life expectancy
* HIV negative
* Not pregnant or nursing

PRIOR CONCURRENT THERAPY:

Biologic therapy

* Not specified

Chemotherapy

* Not specified

Endocrine therapy

* Not specified

Radiotherapy

* Not specified

Surgery

* Not specified

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2001-02; Study Completion 2007-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: H. Joachim Deeg, MD, Study Chair — Fred Hutchinson Cancer Center
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States